CLINICAL TRIAL: NCT02128672
Title: Extraforaminal Spinal Stimulation Compared to Conventional Spinal Cord Stimulation to Treat Axial Low Back Pain-A Pilot Study
Brief Title: Spinal Stimulation to Treat Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped because of competing studies
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tim J. Lamer, M.D., Associate Professor of Anesthesiology, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-003985
Record Dates: First submitted 2014-02-18; First posted 2014-05-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain; Lumbar Back Pain; Lumbago
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional SCS lead (Active Comparator): Conventional Thoracic-lumbar SCS lead placement
  Interventions: Procedure: Spinal Cord Stimulator Lead Placement
- SCS Experimental Lead Placement (Experimental): Experimental SCS lead placement in a novel position
  Interventions: Procedure: Spinal Cord Stimulator Lead Placement

INTERVENTIONS:
Procedure: Spinal Cord Stimulator Lead Placement

SUMMARY:
Spinal cord stimulation (SCS) has been used for almost 30 years to treat many intractable back pain conditions. It has demonstrated efficacy in the co-called Failed Back Surgery Syndrome (FBSS) and a recent randomized controlled trial demonstrated significant superiority of SCS over conventional medical therapy to treat patients with FBSS. Another trial has demonstrated superiority of SCS over repeat surgery in the same patient population. However, the ability to reliably capture the low back with paresthesia coverage has remained challenging and elusive despite numerous strategies designed to overcome this limitation. Strategies that have been introduced but so far with limited success include transverse multiple lead stimulation, high frequency stimulation, peripheral field stimulation, and dorsal root ganglion (DRG) stimulation. To date, none of these strategies have been able to reliably overcome the long-term problems of paresthesia capture and pain relief of the low back.

This proposal describes a new spinal stimulation technique designed to improve the likelihood of low back stimulation by targeting the nerve supply to the two most commonly affected pain producing structures in the back, the facet joints and the intervertebral disks. The technique has proven to be feasible in a cadaver model with ease of lead placement at the desired targets

ELIGIBILITY:
Inclusion:

* Patients with one sided low back pain
* Failed standard conservative care including medications, physical therapy, and/or injections
* Pain greater than 6 months

Exclusion:

* Pregnancy
* Previous spine surgery
* Pain radiating beyond/below the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Did the participant have paresthesia coverage from the stimulation? | Baseline to 4 days
  This is a simple yes or no outcome. Either the patient is able to feel the stimulation paresthesia in the area of his or her back where he or she has pain (outcome is yes) or they do not feel it (outcome is no).

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NRS) | Baseline to 4 days
  NRS is a validated back pain outcome scale
Patient preferred stimulation-Likert Scale | baseline to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Tim Lamer, MD, Principal Investigator — Mayo Clinic